CLINICAL TRIAL: NCT05548868
Title: Feasibility Testing and Pilot RCT of Eating for Wellness (E4W) - An Image-Recognition Dietary Assessment App for Use in Adolescents With Obesity
Brief Title: Pilot RCT of E4W App in Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Jill Hamilton, Division Head, Endocrinology, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1000079525
Record Dates: First submitted 2022-09-12; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Pediatric Obesity
Keywords: Pediatric Obesity; Weight management; Dietary Assessment; Digital health applications; Adolescents; Mobile health
MeSH Terms: conditions — Pediatric Obesity | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Open-label, parallel groups, pilot randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): Patients will receive standard dietary counselling and use of E4W mobile app
  Interventions: Device: E4W mobile app; Behavioral: Standard Care
- Control Arm (Active Comparator): Patients will receive standard dietary counselling. No use of E4W.
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Device: E4W mobile app — Eating for Wellness (E4W) is a mobile application that analyzes photos of meals taken by the user and determines the nutritional profile. Nutritional content is then directly transmitted to the dietitian.
  Arms: Experimental Arm
Behavioral: Standard Care — Patients will receive standard dietary counselling as part of the weight management program.

SUMMARY:
Recommendations for weight management in adolescents with obesity include setting small goals to improve eating behaviours. This frequently includes manually recording food intake over a few days. This is particularly challenging for adolescents as they do not enjoy writing down what they eat, leading to incomplete records. To address this, mobile applications (apps) can easily capture what is eaten through photos. Eating for wellness (E4W) is an app that analyzes photos of meals taken by the user and determines the nutritional profile. The investigators will conduct a pilot randomized controlled trial to determine whether E4W can be implemented successfully and its preliminary effectiveness and impact on dietary intake in adolescents with obesity participating in SickKids' weight management program.

DETAILED DESCRIPTION:
Adolescents are at increased susceptibility for developing obesity-related health issues, with poor eating patterns and increased sedentary behaviours. Recommendations for pediatric obesity management include frequent dietary assessments with health care providers. However, youth often avoid logging their dietary intake through traditional methods. To address this need, image-based mobile applications (apps) are emerging as tools for assessing intake and enhancing participant engagement in weight management programs. However, limited research has been done to characterize eating patterns and diet quality using nutrition smartphone apps in this population. In this study, the investigators will use Eating for Wellness (E4W), an app that analyzes photos of meals taken by the user and determines the nutritional profile. Nutritional content is directly transmitted to the dietitian and remains invisible to the user. E4W provides adolescents with feedback, goal-setting, and tailored support from their dietitian.

The objective of this proposal is to determine whether E4W can be implemented successfully and its preliminary effectiveness and impact on dietary intake in adolescents with obesity participating in a weight management program. The study population will consist of adolescents in the weight management program without an eating disorder, who have the ability to use a smartphone.

Adolescents will be randomly placed in a control (standard care plus logging with default phone camera app only) or experimental group (standard care plus E4W) for 4 weeks. The investigators will assess feasibility and preliminary effectiveness of E4W in improving dietary intake in adolescents with obesity.

Ultimately, our results will inform the design of a larger randomized controlled trial to assess E4W's suitability in replacing current tools for dietary assessment in adolescents with obesity and other populations of children where dietary assessment is important.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in pediatric weight management program
* BMI > or equal to 97th percentile for age and sex
* English-speaking
* Own a smartphone

Exclusion Criteria:

* Non-English speaking
* Severe cognitive impairments that could preclude assessment
* Undergone bariatric surgery
* Diagnosed eating disorder

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-08-05 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Implementation - Accrual Rate | Week 4
  Accrual rate (number of patients who completed the trial) will be tracked to determine feasibility of implementation
Feasibility of Implementation - Technical difficulties | Week 4
  Technical difficulties (total number of technical difficulties encountered) will be tracked to determine feasibility of implementation
Feasibility of Implementation - Patient Satisfaction | Week 4
  Patient Satisfaction (measured using Acceptability E-Scale)

SECONDARY OUTCOMES:
Change in dietary intake | Week 4
  To examine preliminary effectiveness of E4W, overall change in dietary intake and achievement of goals will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Jill Hamilton, MD, MSc, Principal Investigator — Division Head of Endocrinology
Locations (1):
- SickKids, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oei K, Choi EE, Bar-Dayan A, Stinson JN, Palmert MR, Alfonsi JE, Hamilton J. An Image-Recognition Dietary Assessment App for Adolescents With Obesity: Pilot Randomized Controlled Trial. JMIR Form Res. 2024 Dec 2;8:e58682. doi: 10.2196/58682. PMID 39621405